CLINICAL TRIAL: NCT00259831
Title: Efficacy of Cold-FX (CVT-E002) in the Prevention of Upper Respiratory Tract Infections in Healthy Adult Employees in Continuing Care Facilities
Brief Title: Efficacy of Cold-FX (CVT-E002) in the Prevention of Upper Respiratory Tract Infections in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CV Technologies (Industry)
Collaborators: Capital Health, Canada (Other)
Organization: Afexa Life Sciences Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CVT-E002-2005-3
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Upper Respiratory Infection
Keywords: cold; influenza
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold; Influenza, Human | interventions — COLD-fX

INTERVENTIONS:
Drug: CVT-E002 (Cold-FX); a natural health product

SUMMARY:
The purpose of the Study is to determine the prophylactic effects of CVT-E002 treatment for upper respiratory tract infections in healthy adult employees working with residents in continuing care facilities. It is hypothesized that the use of CVT-E002 will effectively reduce the incidence, severity and duration of upper respiratory infections among the participants when compared to placebo.

DETAILED DESCRIPTION:
Eligible continuing care employees will be randomly assigned to either the treatment or placebo group with equal numbers in each group. The treatment will consist of taking two capsules of CVT-E002 (400mg)or placebo every morning, after breakfast, for a period of 12 weeks. The subjects will be given an assessment form to log specific symptoms on a daily basis if they get a cold.

Symptoms include sore throat, runny nose, nasal congestion, hoarseness, cough, earaches, and fever. Subjects will be required to maintain the same dosing even during an upper respiratory infection and will be requested not to take any additional medication for their upper respiratory infection unless prescribed by their family physicians.

ELIGIBILITY:
Inclusion Criteria:

* age 18-64 years
* not pregnant or breast feeding
* good general health

Exclusion Criteria:

* medical conditions: HIV infection; malignancy; cardiovascular disease; hypertension; renal, pulmonary or hepatic abnormalities; neurologic or psychiatric disease; tuberculosis; multiple sclerosis; recent acute respiratory infection (<2 weeks)
* medications: warfarin; immunosuppressive therapy; corticosteroids; phenalzine; pentobarbital; haloperidol
* major surgical procedure in the previous six months
* history of alcohol/drug abuse
* pregnancy and lactation in women

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500
Dates: Start 2005-12; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of CVT-E002 in reducing the number of upper respiratory infections during the study.

SECONDARY OUTCOMES:
To test if the prophylactic management with CVT-E002 decreases the severity and duration of symptoms related to an upper respiratory tract infection.

CONTACTS AND LOCATIONS:
Overall Officials: Gerry Predy, MD, Principal Investigator — Capital Health, Canada
Locations (1):
- The Capital Care Group Continuing Care facilities, Edmonton, Alberta, Canada